CLINICAL TRIAL: NCT00622934
Title: Relationship Between Clinical Recovery and Oxidative Stress and Inflammation Following Usage of Erythropoietin in Admitted Traumatic Patient In Intensive Care Unit
Brief Title: Relationship Between Erythropoietin Administration and Stress Responses in Trauma Patients
Acronym: EPREX
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Pharmaceutical Sciences Research Center Tehran University of Medical SCIENCES, Pharmaceutical Sciences Research Center Tehran University of Medical SCIENCES
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 425/195 13/4/86
Record Dates: First submitted 2008-02-13; First posted 2008-02-25 (Estimated); Last update posted 2010-11-18 (Estimated); Status verified 2010-11

CONDITIONS: Multiple Trauma
Keywords: multiple trauma
MeSH Terms: conditions — Multiple Trauma | interventions — Erythropoietin; Epoetin Alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: erythropoietin
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: erythropoietin — 300mg/kg erythropoietin 3 times on the first week of admission
  Other Names: EPREX
  Arms: 1
Drug: placebo — placebo
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether Erythropoietin decrease stress responses and inflammation in trauma patient.

DETAILED DESCRIPTION:
Transfusion of blood products has many disadvantages. Erythropoietin is used to increase red blood cells production and decrease such disadvantages.In some studies anti inflammatory effects is shown for Erythropoietin.

One of the most problems in the intensive care unit is stress response. we are going to evaluate effects of erythropoietin on oxidative stress and inflammation in trauma patient in intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* All multiple trauma patients>16 years with informed consent

Exclusion Criteria:

* Hypertension
* Allergy
* Erythroid leukemia
* Pregnancy and breast feeding
* Pre operative patient
* Severe cardiovascular and cerebrovascular diseases
* Thromboembolic disorders

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-07; Primary Completion 2008-05 (Estimated); Study Completion 2008-05 (Estimated)

PRIMARY OUTCOMES:
apachi 2 saps 30 days mortality | untill discharge

SECONDARY OUTCOMES:
30 days mortality | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: MOJTABA MOJTAHEDZADE, Study Chair — TUMS; MOSTAFA MOHAMMADY, Principal Investigator — TUMS; MOJTABA MOJTAHED, Study Director — TUMS
Locations (1):
- Sina Hospital, Tehran, Iran